CLINICAL TRIAL: NCT06788691
Title: Efficacy of Luspatercept In Clonal Cytopenias of Uncertain Significance
Brief Title: Luspatercept for Clonal Cytopenias of Uncertain Significance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-06027622
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: CCUS Clonal Cytopenia of Undetermined Significance; Anemia; Leukopenia; Thrombocytopenia; Neutropenia
MeSH Terms: conditions — Anemia; Leukopenia; Thrombocytopenia; Neutropenia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Luspatercept (Experimental): Luspatercept administered at 1 mg/kg IV once every 3 weeks
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Administered at 1 mg/kg once every 3 weeks

SUMMARY:
The purpose of this clinical trial is to test how well the drug luspatercept works in improving low blood cell counts in people with clonal cytopenias of uncertain significance (CCUS). The main questions the study seeks to answer include:

* How many patients experience improvements in their low blood counts (red cells, platelets, or white cells) within 24 weeks, based on specific criteria for blood conditions like myelodysplastic syndromes (MDS)?
* How long these improvements last before the condition worsens or changes.
* The percentage of participants showing improvements at 12, 24, and 48 weeks.
* How long it takes for the condition to progress to more severe diseases like myeloid disorders.
* How long red blood cell responses last and how quickly these responses are seen.
* The average change in hemoglobin levels over 24 weeks.
* How many patients need blood transfusions during the study and how soon transfusions are required.
* Changes in participants' well-being and energy levels based on a standardized questionnaire.
* Monitoring for any side effects, including progression to MDS or leukemia, heart-related issues, or sudden increases in hemoglobin.

Participants will:

* Receive luspatercept as an injection every three weeks.
* Visit the clinic every three weeks for treatment and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Documentation of a CCUS diagnosis.

  * Clonal cytopenia of undetermined significance (CCUS) is defined as clonal hematopoiesis of indeterminate potential (CHIP) detected in the presence of one or more persistent cytopenias that are otherwise unexplained by hematologic or non-hematologic conditions and that do not meet diagnostic criteria for defined myeloid neoplasms. Cytopenia definitions for diagnosis of CCUS include Hb <13 g/dL in males and <12 g/dL in females for anemia, absolute neutrophil count <1.8 ×109/L for leukopenia, and platelets <150 × 109/L for thrombocytopenia.
  * Patients should harbor somatic mutations of myeloid malignancy-associated genes detected in the blood or bone marrow at a variant allele fraction (VAF) of ≥ 2% (≥4% for X-linked gene mutations in males
* Clinically significant cytopenias demonstrated in two separate lab draws 3 months apart and defined as cytopenia in any one of the following:

  * Anemia: Transfusion dependent (LTD or HTD for Hb < 9 g/dL based on IWG 2018 criteria). Exception for higher threshold up to 10g/dL for documented moderate or severe angina pectoris, cardiac or pulmonary insufficiency, or ischemic neurologic diseases (per IWG 2018 consensus recommendation).
  * Anemia NTD: symptomatic NTD CCUS with Hb <10 g/dl, symptomatic defined as moderate or worse on ≥ 1 Patient Global Impression of Severity (PGI-S) item (fatigue, shortness of breath, weakness, or dizziness)
  * Thrombocytopenia: platelet count less than 30,000 /microL or < 50,000/microL with documented bleeding events or high risk for bleeding, for example on blood thinners or drugs that inhibit platelet function for other comorbidities.
  * Neutropenia: Neutropenia below 750/microl are included in the study. For subjects with neutropenia between 750-1000/microl, subjects should have neutropenia AND a history of serious infection(s).
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Adequate organ function as defined by:

  * Direct bilirubin < 3 x ULN. Indirect hyperbilirubinemia from hemolysis or Gilberts disease are not considered as impaired.
  * Estimated Creatinine clearance >30 ml/min by institutional standard (either MDRD or Cockcroft Gault or measured by 24 hour urine clearance.
  * ALT and AST < 3 x ULN
* Females of childbearing potential (FCBP), defined as a sexually mature woman who: 1) has achieved menarche at some point, 2) not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or amenorrhea due to other medical reasons does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), must:

  * Have two negative pregnancy tests (serum or urine) as verified by the investigator prior to starting study therapy (unless the screening pregnancy test was done within 72 hours of W1D1). She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment.
  * Either commit to true abstinence1 from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, highly effective contraception2 without interruption, 5 weeks prior to starting investigational product, during the study therapy (including dose interruptions), and for 12 weeks after discontinuation of study therapy.

Male subjects must:

- Practice true abstinence1(which must be reviewed prior to each IP administration or on a monthly basis [e.g., in the event of dose delays]) or agree to use a condom (latex or non-latex, but not made out of natural [animal] membrane) during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks following investigational product discontinuation, even if he has undergone a successful vasectomy.

Contraception

* True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception].
* Highly effective contraception is defined in this protocol as the following (information will also appear in the ICF): Hormonal contraception (for example, birth control pills, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation (tying your tubes); or a partner with a successful vasectomy.

Exclusion Criteria:

* Concurrent malignancy requiring active systemic therapy
* Diagnosis of MDS, AML, MPN or any other myeloid malignancy in the patient's lifetime
* Active uncontrolled infection that in the investigators opinion will affect study procedures and/or results
* Active uncontrolled hypertension not responding to blood pressure lowering medications which in the investigator's opinion will be harmful for the patient.
* Use of ESA or growth factors within four weeks prior to the start of the study
* Known risk factors for thromboembolism (splenectomy, concomitant use of hormone replacement therapy or recent uncontrolled pulmonary embolism or DVT in the last 6 months). Subjects adequately controlled on anticoagulation are permitted.
* Pregnant or nursing women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of study treatment and for up to 130 days after last dose of study drug. Basic contraception methods are defined in Section 4.4.

  * Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (i.e. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks prior to first dose of study drug. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of childbearing potential. If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the Informed Consent Form (ICF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients achieving cytopenia responses as defined by HI-E, HI-P, HI-N, mHI-E responses | 24 Weeks
  Adapted from International Working Group (IWG) 2018 response definition for Myelodysplastic Syndromes

SECONDARY OUTCOMES:
Duration of cytopenia response | 24 Weeks
  The duration of cytopenia response, defined as the time from the first documented achievement of cytopenia response to the loss of response or disease progression.
Percentage of Participants Achieving Hematologic Response | 12 Weeks
Percentage of Participants Achieving Hematologic Response | 24 Weeks
Percentage of Participants Achieving Hematologic Response | 48 Weeks
Time to Transformation to Myeloid Disease | Week 4 (Cycle 1 Week 1) to 24 Weeks
  Time to transformation to myeloid disease as evidenced by bone marrow morphology findings.
Duration of modified hematologic improvement-erythroid (mHI-E) | Week 4 (Cycle 1 Week 1) to 24 Weeks
  Duration of modified hematologic improvement-erythroid (HI-E) per IWG 2006
Time to mHI-E | Week 4 (Cycle 1 Week 1) to 24 Weeks
  Time to hematologic improvement-erythroid (mHI-E) per IWG 2006
Mean Change Hemoglobin (Hb) | Baseline, 24 Weeks
Number of Patients Converting to Transfusion Dependence (TD) | 12 Weeks
  Number of patients who convert to transfusion dependence (≥ 3 units/16 weeks per IWG 2018 criteria) at 12 weeks, provided they were not transfusion-dependent at study entry.
Number of Patients Converting to Transfusion Dependence (TD) | 24 Weeks
  Number of patients who convert to transfusion dependence (≥ 3 units/16 weeks per IWG 2018 criteria) at 24 weeks, provided they were not transfusion-dependent at study entry.
Number of Patients Converting to Transfusion Dependence (TD) | 48 Weeks
  Number of patients who convert to transfusion dependence (≥ 3 units/16 weeks per IWG 2018 criteria) at 48 weeks, provided they were not transfusion-dependent at study entry.
Time to the first red blood cell transfusion | 24 Weeks
Mean Change in FACT-An Total Scores | Baseline, 24 Weeks
  Functional Assessment of Cancer Therapy-Anemia (FACT-An) total scores. The FACT-An (Functional Assessment of Chronic Illness Therapy - Anemia) questionnaire is a validated tool designed to evaluate the quality of life in patients with anemia, especially those receiving treatment for cancer-related anemia. The total FACT-An score ranges from 0 to 188.
Mean Change in FACT-An Subscale Scores | Baseline, 24 Weeks
  Functional Assessment of Cancer Therapy-Anemia (FACT-An) subscale scores. The FACT-An (Functional Assessment of Chronic Illness Therapy - Anemia) questionnaire is a validated tool designed to evaluate the quality of life in patients with anemia, especially those receiving treatment for cancer-related anemia. The questionnaire consists of five subscales, with score ranges varying by subscale: 0-28, 0-24, or 0-80.
Safety as assessed by number of subjects with MDS/AML progression | Week 4 (Cycle 1 Week 1) to 24 Weeks
Safety as assessed by number of cardiovascular events | Week 4 (Cycle 1 Week 1) to 24 Weeks
Safety as assessed by number of subjects with rapid hemoglobin rise | Week 4 (Cycle 1 Week 1) to 24 Weeks
Number of participants achieving Red Blood Cell Transfusion Independence (RBC-TI) for at least 24 consecutive weeks | Week 4 (Cycle 1 Week 1) to 24 Weeks
Number of participants achieving Hematologic Improvement-Erythroid (HI-E) for at least 24 consecutive week as per IWG 2006 criteria. | Week 4 (Cycle 1 Week 1) to 24 Weeks
Duration of RBC-TI greater than 16 Weeks | Week 1 to Week 24
  Duration of red blood cell transfusion independence (RBC-TI) for greater than 16 weeks
Number of participants achieving RBC-TI | 16 Weeks
  Number of participants achieving RBC-TI over 16 weeks along with a mean hemoglobin increase of >1.5 g/dL over the same time period.
Change in cardiac biomarkers over the treatment period | Baseline, 24 Weeks
Mean Change Health-related quality of life (HRQoL) Assessment | 12 Weeks
  The Functional Assessment of Cancer Therapy - Anemia (FACT-An) is the Health-Related Quality of Life (HRQoL) tool used in this study. The lowest possible score is 0, which reflects the worst possible quality of life, indicating severe impairments in overall well-being and significant anemia-related symptoms. The highest possible score is 188, representing the best possible quality of life, with minimal or no symptoms and optimal functioning across all domains, including anemia-related concerns.
Mean Change Health-related quality of life (HRQoL) Assessment | 24 Weeks
  The Functional Assessment of Cancer Therapy - Anemia (FACT-An) is the Health-Related Quality of Life (HRQoL) tool used in this study. The lowest possible score is 0, which reflects the worst possible quality of life, indicating severe impairments in overall well-being and significant anemia-related symptoms. The highest possible score is 188, representing the best possible quality of life, with minimal or no symptoms and optimal functioning across all domains, including anemia-related concerns.
Mean Change Health-related quality of life (HRQoL) Assessment | 48 Weeks
  The Functional Assessment of Cancer Therapy - Anemia (FACT-An) is the Health-Related Quality of Life (HRQoL) tool used in this study. The lowest possible score is 0, which reflects the worst possible quality of life, indicating severe impairments in overall well-being and significant anemia-related symptoms. The highest possible score is 188, representing the best possible quality of life, with minimal or no symptoms and optimal functioning across all domains, including anemia-related concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Pinkal Desai, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No